CLINICAL TRIAL: NCT04763733
Title: Prognostic Scoring System of Laparoscopic Splenectomy in Children With Benign Hematological Diseases.
Brief Title: Laparoscopic Splenectomy in Children
Acronym: splenectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, assistant professor of pediatric surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 33872/6/20
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Laparoscopic Splenectomy; Children; Benign Blood Diseases
Keywords: laparoscopic splenectomy,; children; prognostic score; benign hematological diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | Pediatric Postmarket Surveillance: Yes

INTERVENTIONS:
Other: laparoscopic splenectomy — surgical

SUMMARY:
Laparoscopic splenectomy (LS) gained popularity since it has been described for the first-time during nineties of past century. It has become "golden method" for splenectomy in all ages including children

DETAILED DESCRIPTION:
Background: laparoscopic splenectomy (LS) gained popularity during the last years in pediatric age group. Benign hematological diseases represent the main indications of that procedure. There are some score systems of difficulty of the technique but they are for adult patients. The aim is to develop a prognostic score system of LS in children with benign hematological diseases.

Methods: LS was performed in all children with benign hematological diseases. LS was done by the same team. They operated children in lateral decubitus position. The control of pedicle was achieved using bipolar sealing devices, polymer clips or endoscopic linear staplers. Preoperative, operative, and postoperative data were recorded and analyzed. Children were divided into two groups A and B according to the development of complications.

ELIGIBILITY:
Inclusion Criteria:

* children with benign hematological diseases

Exclusion Criteria:

* malignant hematological diseases

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
prognosis of procedure | from day 0 to 7 days
  number of patients with peritoneal collections, number of patients having pancreatitis, number of patients staying more than two days postoperative

IPD SHARING:
Plan to Share IPD: No